CLINICAL TRIAL: NCT04090567
Title: Overcoming PARP Inhibitor Resistance in BRCA Germline Mutation Positive Advanced Breast Cancer
Brief Title: Olaparib With Cediranib or AZD6738 for the Treatment of Advanced or Metastatic Germline BRCA Mutated Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0062; NCI-2019-04148 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0062 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-08-22; First posted 2019-09-16 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Advanced Breast Carcinoma; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Germline BRCA1 Gene Mutation; Germline BRCA2 Gene Mutation; HER2/Neu Negative; Metastatic Breast Carcinoma; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms | interventions — cediranib; ceralasertib; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (olaparib plus cediranib) (Experimental): Patients receive olaparib PO BID and cediranib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cediranib; Drug: Olaparib
- Arm II (olaparib plus ceralasertib) (Experimental): Patients receive olaparib PO BID on days 1-28 and ceralasertib PO QD on days 1-7. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ceralasertib; Drug: Olaparib

INTERVENTIONS:
Drug: Cediranib — Given PO
  Other Names: AZD2171
  Arms: Arm I (olaparib plus cediranib)
Drug: Ceralasertib — Given PO
  Other Names: AZD6738
  Arms: Arm II (olaparib plus ceralasertib)
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281

SUMMARY:
This phase II trial studies how well olaparib with cediranib or AZD6738 works in treating patients with germline BRCA mutated breast cancer that has spread to other places in the body (advanced or metastatic). Olaparib, cediranib, and AZD6738 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the objective response rate (ORR) of olaparib plus cediranib and olaparib plus ceralasertib (AZD6738) combinations in patients with advanced or metastatic breast cancer with germline BRCA (breast cancer susceptibility gene) mutations who have been previously treated with PARP inhibitors.

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of olaparib in combination with cediranib and in combination with AZD6738 in patients with advanced or metastatic breast cancer with germline BRCA mutations.

II. To assess duration of response (DOR) to treatment. III. To assess best response. IV. To estimate progression free survival (PFS).

EXPLORATORY OBJECTIVES:

I. To evaluate BRCA1 expression at baseline and on progression. II. To evaluate hypoxia markers at baseline and on progression. III. To evaluate levels of angiogenesis/ inflammatory markers including VEGF (vascular endothelial growth factor) at baseline and on progression.

IV. To evaluate novel markers of resistance and response to PARP inhibitor in baseline and upon progression of disease in tumor tissue that are identified by the investigator's basic science collaborator's ongoing studies in vitro and in vivo.

V. To evaluate circulating tumor deoxyribonucleic acid (DNA) at baseline and on progression.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive olaparib orally (PO) twice daily (BID) and cediranib PO once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive olaparib PO BID on days 1-28 and ceralasertib PO QD on days 1-7. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Women age greater than 18 years with advanced/metastatic HER2 negative, BRCA germline positive breast cancer. Estrogen receptor positive (ER+) patients must have progressed on a prior endocrine therapy or are considered inappropriate for any FDA approved endocrine therapies for ER+ breast cancer.
3. Eligible patients must agree to a mandatory fresh biopsy (excluding bone) at screening. In addition, if available, an archival tissue sample will also be collected at screening.
4. Patients must have normal organ and bone marrow function measured within 28 days (baseline screening) as defined below:

   * Hemoglobin (Hgb) >/= 10.0 g/dL with no blood transfusion in the past 28 days prior to the administration
   * Absolute neutrophil count (ANC) >/= 1.5 x 109/L with no GCSF administration within 28 days prior to administration of study treatment
   * Platelet count >/= 100 x 109/L
   * Total bilirubin </= 1.5 x institutional upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) / Alanine aminotransferase (ALT) </=3.0 x institutional upper limit of normal unless liver metastases are present in which case they must be </=5x ULN

4) Eastern Cooperative Oncology Group (ECOG) performance status 0-1 5) Patients must have life expectancy >/= 16 weeks. 6) Negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on Cycle 1 day 1 and during the study for child bearing potential women.

• Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥ 60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry and be using highly effective contraception (that is, methods with a failure rate of less than 1% per year) for both male and female subjects if the risk of conception exists (Note: The effects of the trial treatment on the developing human fetus are unknown; thus, women of childbearing potential and men must agree to use highly effective contraception, defined in Appendix E or as stipulated in national or local guidelines). Highly effective contraception must be used 30 days prior to first trial treatment administration, for the duration of trial treatment, and at least for 1 month after stopping trial treatment.

7) Patients is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations. 8) Patient has measurable disease, per RECIST v 1.1. At least one lesion, not previously irradiated or biopsied for this study that can be accurately measured at baseline as >/= 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI).

9) Willingness to undergo baseline biopsy of metastatic lesion (repeat biopsy at progression/or end of the study is optional) 10) Willingness to have research blood draw at baseline and at progression/end of the study 11) Patient should have previously treated with any PARP inhibitor ((neo)adjuvant or metastatic) setting) and must have remained on treatment for >/= 2 months prior to progression of disease.

12) Able to swallow and retain oral medications and without gastrointestinal (GI) illnesses that would preclude absorption of Olaparib or ceralasertib.

13) Non-english speaking subject can be enrolled

Exclusion Criteria:

1. Patients who have had chemotherapy or RT within 3 weeks ( or less than 1 week if on weekly chemotherapy) prior to start of the study agents. or persisting >/= Grade 2 CTCAE toxicity (except alopecia and Grade 2 peripheral neuropathy) from previous anti-cancer treatment(s), or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier. No washout time period is needed for PARP inhibitors.
2. Patients received any other investigational agents within the past 4 weeks.
3. Patients with untreated brain metastases, spinal cord compression, or evidence of symptomatic brain metastases or leptomeningeal disease as noted on computed tomography (CT) or magnetic resonance imaging (MRI) scans should be excluded from this clinical trial. Patient with known and treated brain metastases is allowed in this study if they fulfil the following criteria: The lesions have improved or remained stable radiographically and clinically for at least 6 weeks after completion of brain irradiation or stereotactic brain radiosurgery. Patients can be on steroids not more than 10 mg/day if started 4 weeks prior to initiation of study drug).
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Olaparib or ceralasertib.
5. Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 (See Appendix A) are ineligible, unless discontinues within the washout period (2 weeks for CYP3A4 inhibitors and 4weeks for CYP3A4 inducers) as described in Appendix A. Dihydropyridine calcium-channel blockers are permitted for management of hypertension. Other medications described in Appendix A should be discontinued within the washout period prior to the initiation of study drugs. In addition, patients enrolled in Olaparib+ ceralasertib arm, co-administration of study drug with substrates of OATP1B1 and Pgp (P-glycoprotein) inhibitor or inducer is prohibited.
6. Current use of natural herbal products (see Appendix A) or other complementary alternative medications (CAM) or "folk remedies" should be discontinued 7 days prior to the initiation of study drugs.

8) Patients with concomitant or prior invasive malignancies within the past 5 years. Subjects with treated limited stage basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the breast or cervix are eligible.

9) Uncontrolled inter-current illness including, but not limited to, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.

10) History of myocardial infarction, stroke or transient ischemic attack within 6-12 months. Current condition requiring concurrent use of drugs or biologics with anti-arrhythmic or proarrhythmic potential 11) History of hypertensive crisis or hypertensive encephalopathy within 3 years.

12) Clinically significant peripheral vascular disease or vascular disease (abdominal aortic aneurysm (>5cm) or aortic dissection). If known history of abdominal aortic aneurysmwith

* 4cm in diameter, all the following criteria must be met:

  * An ultrasound (US) within the last 6 months will be required to document that it is </= 5cm
  * Patient must be asymptomatic from the aneurysm.

    13) A major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to starting study drug (percutaneous/endobronchial biopsies are allowed). The patient must have recovered from any effects of any major surgery and surgical wound should have healed prior to starting treatment.

    14) Patients may not have current signs and/or symptoms of bowel obstruction within 3 months prior to starting study drugs, except if it was a temporary incident (improved within < 24hrs with medical management).

    15)History of haemoptysis or any significant bleeding within the last 1 month prior to enrolment. 16) Presence of cavitation of central pulmonary lesion 17) Intra-abdominal abscess within the 3 months prior to enrolment. Patient with history of GI perforation. History of abdominal fistula will be considered eligible, if the fistula was surgically repaired, there has been no evidence of fistula for at least 6 months prior to starting treatment, and patient is deemed to be at low risk of recurrent fistula.

    18) Patients may have current dependency on IV hydration or total parenteral nutrition (TPN).

    19) Patients may have features suggestive of myelodysplastic syndrome (MDS) or acute myelogenous leukemia (AML) on peripheral blood smear or bone marrow biopsy, if clinically indicated. 20) As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases, active bleeding diatheses, renal transplant, or active infection including any patient known to have hepatitis B, hepatitis C and human immunodeficiency virus (HIV).

Screening for chronic conditions is not required 21) Any condition that, in the opinion of the treating investigator would interfere with evaluation of the investigational product or interpretation of subject safety or study results.

22) Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.

23) Prior exposure to Ceralasertib 24) Patients with uncontrolled seizure 25) Any of the following cardiac criteria:

* Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >450 milli-second, or patients with congenital long QT syndrome or family history of unexplained sudden death under 40 years of age
* Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block).

  26) Patients at risk of brain perfusion problems, e.g., carotid stenosis 27) Patients with relative hypotension (< 100/60 mm Hg) or clinically relevant orthostatic hypotension (>/= 20 beats per minute change in pulse including a fall in blood pressure of

  >/=20mm Hg associated with dizziness, syncope, and blurred vision, from lying down or sitting to standing). Uncontrolled hypertension requiring clinical intervention.

  28) Breast feeding/lactating/pregnant women. 29) Prior allogeneic bone marrow transplant or double umbilical cord blood transplantation.

  30) A diagnosis of ataxia telangiectasia 31) Major surgery within 3 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 30 days post treatment
  Defined as proportion of patients with reduction in tumor burden (complete response [CR] or partial response [PR] as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. The exact two-sided 95% confidence interval for the ORR will be reported.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 30 days post treatment
  PFS will be estimated using the Kaplan-Meier method with the 95% confidence intervals (CIs). Will analyze aggregate data from selected arms of the trial using Cox proportional hazards and logistic regression to identify study factors related to outcomes including response and PFS. Hazard ratios and odds ratios with their 95% confidence intervals and p-values will be reported. Model assumptions will be verified.
Duration of response (DOR) | Up to 30 days post treatment
  DOR will be estimated using the Kaplan-Meier method with the 95% CIs. Will analyze aggregate data from selected arms of the trial using Cox proportional hazards and logistic regression to identify study factors related to outcomes including response and PFS. Hazard ratios and odds ratios with their 95% confidence intervals and p-values will be reported. Model assumptions will be verified.

OTHER OUTCOMES:
Biomarker analysis | Up to 30 days post treatment
  Will be done using Fisher's exact tests, Mann-Whitney U tests or McNemar's test will be applied depending the type of data we observe. For the pre- and post- therapy biomarker and outcome analysis, paired t- test or Wilcoxon signed-rank will be applied for the continuous variables. McNemar's test will be applied for categorical variables. Fisher's exact test will be applied for the association between hypoxia positivity and objective response. Will use this information to estimate the 95% confidence intervals for future pivotal trials.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Arun, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org